CLINICAL TRIAL: NCT04014608
Title: Admission Toxigenic C. Difficile Surveillance to Reduce Hospital Onset C. Difficile Infection (CDI)
Brief Title: Protocol for Admission Toxigenic C. Difficile Surveillance
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Other Study IDs: QAInitiative6.18.2016
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile Infection; Infection Control; Quality Improvement; Active Surveillance testing
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baseline Control: Standard Practice before the intervention was introduced
  Interventions: Other: Standard Practice to Prevent Hospital Onset CDI
- Intervention initiative: Standard Practice plus Admission Surveillance for toxigenic C. difficile.
  Interventions: Other: Standard Practice to Prevent Hospital Onset CDI

INTERVENTIONS:
Other: Standard Practice to Prevent Hospital Onset CDI — Bleach cleaning of rooms, use of required soap/water hand hygiene for CDI patients, hand hygiene monitoring, portable ultraviolet (UV) light room disinfection, and monitoring of room cleaning.

SUMMARY:
Background: Clostridioides (formerly Clostridium) difficile Infection (CDI) is a persistent healthcare issue. In the US, CDI is the most common infectious cause of hospital-onset (HO) diarrhea.

Objective: Assess the impact of admission testing for toxigenic C. difficile colonization on the incidence of clinical disease.

Design: Pragmatic stepped-wedge Infection Control initiative. Setting: NorthShore University HealthSystem (NorthShore) is a four-hospital system near Chicago, Illinois.

Patients: All patients admitted to the four hospitals during the initiative. Interventions: From September 2017 through August 2018 the investigators conducted a quality improvement program where admitted patients had a peri-rectal swab tested for toxigenic C. difficile. All colonized patients were placed in contact precautions.

Measurements: The investigators tested admissions who: i) had been hospitalized within two months, ii) had a past C. difficile positive test, and/or iii) were in a long-term care facility within six months. The investigators measured compliance with all other measures to reduce the incidence of HO-CDI.

Limitations: This was not a randomized controlled trial, and multiple prevention interventions were in place at the time of the admission surveillance initiative.

DETAILED DESCRIPTION:
Background:

Clostridium difficile infection (CDI) remains a constant, even increasing, clinical infection threat in the United States and Europe. New preventive strategies are urgently needed. Current control measures do not target asymptomatic carriers, despite evidence that they can contaminate the hospital environment and health care workers' hands; a risk to potentially transmit C. difficile to other patients. Of special importance is that not only is disease prevalence increasing, but severity of illness and mortality also is on the rise. The investigators have implemented many interventions at our healthcare system including bleach cleaning of rooms with CDI patients, monitoring of environmental services' room cleaning, hand hygiene education and even UV light disinfection of rooms harboring CDI patients, and none have been consistently effective. The investigators believe that CDI is much like methicillin resistant Staphylococcus aureus (MRSA), in that many more patients are colonized than infected, and one (perhaps the optimal) way to curtail disease is to interrupt transmission by identifying carriers and placing them into contact (glove and gown) precautions.

The investigators propose to test this hypothesis with a quality improvement program study at NorthShore. The primary goal is to demonstrate that surveillance testing for C. difficile colonization at the time of admission and contact precaution isolation of those positive will reduce spread of the organism as well as lower clinical CDI. The investigators secondary goals are to demonstrate a reduction in C. difficile infection incidence after implementation of this program and demonstrate that such a program is cost effective.

Study Methods:

We have collected CDI disease rates for 10 years. One of our hospitals admits a high number of patients from long term care facilities (LTCFs) and currently has a rate of infection at 11 cases/10,000 patient days, and this facility served as a pilot site in the program initiative. The nosocomial CDI rate at this facility had been rising during the first quarter of 2016. The investigators plan to introduce peri-rectal (intra-anal) swab testing for C. difficile on all admissions accompanied by isolation of positive patients, which the investigators hypothesize will lower the rate to 3 cases/10,000 patient days. In absolute numbers, the goal is to reduce the rate from 4 nosocomial cases per month down to 1 nosocomial case per month. This is intended to provide a sample size that can demonstrate a level of significance at p<.05 for disease reduction with the intervention when compared to the same time frame prior to the admission testing intervention.

If the proposed pilot admission screening program is successful, the investigators will show disease is reduced by implementing the admission screening program. At that point, if a successful outcome is achieved, the program will be extended to all 4 hospitals in the NorthShore system.

Additionally, the investigators will be collecting a double headed swab (Culturette) on all patients, so those testing positive will have the second swab cultured for C. difficile. The purpose of this is to validate the Roche C. Diff Cobas test as a valid screen testing platform.

Study Period:

All admissions giving verbal consent to the target pilot hospital will be tested, and the program will continue until at least 2,000 patients have taken part. The admitting nurses or patient care technicians (PCTs) will collect the peri-rectal swab sample specimen. This initial program began on July 1, 2016. The expected primary completion date for the pilot program was December 31, 2016. The complete observation period for the full 4-hospital initiative ended December 31, 2018.

Testing Plan:

Patients admitted to the target hospital will have a peri-rectal swab collected at the time of admission. This will be tested by the Roche cobas C. Diff assay. The investigators will be testing 6 days per week at the central hospital (Evanston Hospital).

Potential Benefit:

A report from Canada (using the BD assay) indicates the concept should work (reference 10 below) - the investigators believe the outcome will be better than or equal to the result of this publication since isolation will include gowns as well as gloves. The investigators will be the first US study to show admission testing works to provide a significant reduction in healthcare-onset C. difficile infection (HO-CDI) and save patient lives.

Initial Supporting References:

1. Dallal RM, Harbrecht BG, Boujoukas AJ, et al. Fulminant Clostridium difficile: an underappreciated and increasing cause of death and complications. Ann Surg 2002;235:363-72.
2. Dubberke ER, Reske KA, Olsen MA, McDonald LC, Fraser VJ. Short- and long-term attributable costs of Clostridium difficile-associated disease in nonsurgical inpatients. Clin Infect Dis 2008;46:497-504.
3. Kuijper EJ, Coignard B, Tull P. Emergence of Clostridium difficile-associated disease in North America and Europe. Clin Microbiol Infect 2006;12 Suppl 6:2-18.
4. Loo VG, Poirier L, Miller MA, et al. A predominantly clonal multi-institutional outbreak of Clostridium difficile-associated diarrhea with high morbidity and mortality. N Engl J Med 2005;353:2442-9.
5. McDonald LC, Owings M, Jernigan DB. Clostridium difficile infection in patients discharged from US short-stay hospitals, 1996-2003. Emerg Infect Dis 2006;12:409-15.
6. Musher DM, Aslam S, Logan N, et al. Relatively poor outcome after treatment of Clostridium difficile colitis with metronidazole. Clin Infect Dis 2005;40:1586-90.
7. Pepin J, Valiquette L, Alary ME, et al. Clostridium difficile-associated diarrhea in a region of Quebec from 1991 to 2003: a changing pattern of disease severity. CMAJ 2004;171:466-72.
8. Zacharioudakis IM, Zervou FN, Pliakos EE, Ziakas PD, Mylonakis E. Colonization with toxinogenic C. difficile upon hospital admission, and risk of infection: a systematic review and meta-analysis. Am J Gastroenterol 2015 Mar;110(3):381-90; quiz 391. doi: 10.1038/ajg.2015.22. Epub 2015 Mar 3.
9. Curry SR, Muto CA, Schlackman JL, Pasculle AW, Shutt KA, Marsh JW, Harrison LH. Use of multilocus variable number of tandem repeats analysis genotyping to determine the role of asymptomatic carriers in Clostridium difficile transmission. Clin Infect Dis 2013 Oct;57(8):1094-102. doi: 10.1093/cid/cit475. Epub 2013 Jul 23.
10. Longtin Y, Paquet-Bolduc B, Gilca R, Garenc C, Fortin E, Longtin J, Trottier S, Gervais P, Roussy JF, Lévesque S, Ben-David D, Cloutier I, Loo VG. Effect of detecting and isolating Clostridium difficile carriers at hospital admission on the incidence of C. difficile infections: A quasi-experimental controlled study. JAMA Intern Med 2016 Apr 25. doi: 10.1001/jamainternmed.2016.0177. [Epub ahead of print]

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission

Exclusion Criteria:

* None

Max Age: 1 Year | Sex: All
Age Groups: Child
Study Population: All patients admitted to NorthShore University HealthSystem comprised of four-hospital system with 789 inpatient beds located north of Chicago, IL.
Sampling Method: Non-Probability Sample
Enrollment: 148549 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Hospital Onset C. difficile Infection | Nine months of a pilot program at one hospital and one year of all 4 hospital application of admission screening
  An altered incidence of this hospital acquired infection

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University HealthSystem Research Institute, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peterson LR, O'Grady S, Keegan M, Fisher A, Zelencik S, Kufner B, Shah M, Lim R, Schora D, Das S, Singh K. Reduced Clostridioides difficile infection in a pragmatic stepped-wedge initiative using admission surveillance to detect colonization. PLoS One. 2020 Mar 19;15(3):e0230475. doi: 10.1371/journal.pone.0230475. eCollection 2020. PMID 32191763